CLINICAL TRIAL: NCT02340507
Title: The Impact of the Glycaemic Index (GI) on Daily Blood Glucose Profiles and Food Intake in Young Chinese Adult Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 2013/00266
Record Dates: First submitted 2015-01-07; First posted 2015-01-16 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes; Obesity; Prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Prediabetic State | interventions — Bread

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High glycemic index (Experimental): The subject will consume a high glycemic index glutinous rice for breakfast (75g available carbohydrates), and a high glycemic index white bread for snack (25g available carbohydrates). The lunch is a standardized, weighed portion buffet.
  Interventions: Other: Rice and bread (high GI)
- Low glycemic index (Experimental): The subject will consume a low glycemic index parboiled basmati rice for breakfast (75g available carbohydrates), and a low glycemic index multigrain bread for snack (25g available carbohydrates). The lunch is a standardized, weighed portion buffet.
  Interventions: Other: Rice and bread (low GI)

INTERVENTIONS:
Other: Rice and bread (high GI) — Rice is a high glycaemic index glutinous rice. Bread is a high glycaemic index white bread.
  Arms: High glycemic index
Other: Rice and bread (low GI) — Rice is a low glycaemic index parboiled basmati rice. Bread is a low glycaemic index multigrain bread.
  Arms: Low glycemic index

SUMMARY:
This study is carried out to find out the inclusion of high and low glycaemic Index (GI) foods to daily meals impact on 24 hour blood glucose fluctuations and food intake.

DETAILED DESCRIPTION:
The GI is a method of classifying foods based on the food's ability to raise the blood glucose level. Low GI foods are recommended as they have a lower impact on blood glucose concentrations and also reduce total food intake. There is very little information on how eating high and low GI foods affect daily blood glucose concentrations in Asians. Therefore, the objective of this study is to observe the effect of eating high and low GI breakfasts and snacks on 24 hour blood glucose concentrations and food consumption in Asian males. Healthy, normal-weight, Chinese males will be recruited. There will be two sessions (consisting of four days for each session) where they will consume either a high or low GI breakfast or snack, and a standardized ad libitum lunch buffet. Their glycaemic response will be measured using a Continuous Glucose Monitoring System (CGMS) throughout the period. The proposed research for the first time demonstrates how the consumption of high and low GI breakfasts and snacks affect subsequent energy intake and 24 hour blood glucose profiles in Asians. These findings will have significant public health benefits for optimum weight and dietary control.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, male
* Age between 21-40 years
* Body mass index between 17 to 24 kg/m2
* Normal blood pressure (120/80 Hgmm)
* Fasting blood glucose < 6 mmol/L

Exclusion Criteria:

* Having any metabolic diseases (such as diabetes, hypertension etc)
* One prescription medication
* Partaking in sports at the competitive and/or endurance levels
* Allergic/intolerant to any of the test foods
* Intentionally restricting food intake
* Smoking

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2014-05 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Glycaemic response (measured 3 hours post consumption using the Continuous Glucose Monitoring System (CGMS) | 3 hours post consumption
  The blood glucose response to low and high GI test foods measured 3 hours post consumption using the Continuous Glucose Monitoring System (CGMS)
Daily blood glucose profile (easured for each low and high GI treatment as the area under the curve over 24 hours using CGMS) | 24 hours
  The daily total blood glucose response is measured for each low and high GI treatment as the area under the curve over 24 hours using CGMS.

SECONDARY OUTCOMES:
Energy intake (The amount of food consumed at the ad libitum lunch is measured by weighed quantities (in grams converted to kilocalories) based on the difference of the weight of food before and after consumption) | Immediately post meal consumption
  The amount of food consumed at the ad libitum lunch is measured by weighed quantities (in grams converted to kilocalories) based on the difference of the weight of food before and after consumption

REFERENCES:
- [Derived] Kaur B, Ranawana V, Teh AL, Henry CJK. The impact of a low glycemic index (GI) breakfast and snack on daily blood glucose profiles and food intake in young Chinese adult males. J Clin Transl Endocrinol. 2015 Jun 11;2(3):92-98. doi: 10.1016/j.jcte.2015.05.002. eCollection 2015 Sep. PMID 29204372